CLINICAL TRIAL: NCT05030337
Title: Does Closed-loop Automated Oxygen Control Reduce the Duration of Mechanical Ventilation? A Randomised Controlled Trial in Ventilated Preterm Infants
Brief Title: Optimising Ventilation in Preterms With Closed-loop Oxygen Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 297749; KCH21-111 (Other: King's College Hospital)
Record Dates: First submitted 2021-08-17; First posted 2021-09-01 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Infant, Premature, Diseases; Airway Morbidity; Mechanical Ventilation Complication
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Intervention Model Description: Participating infants will be randomised either to manual oxygen control or closed-loop automated oxygen control, adjusted by clinical staff as necessary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual oxygen control (No Intervention): Standard ventilation with inspired oxygen concentration adjusted manually as per unit's protocol.
- Closed-loop automated oxygen control (Other): Ventilation with Oxygenie software (closed-loop automated oxygen control system), adjusted by clinical staff as necessary
  Interventions: Device: Closed-loop automated oxygen control (Oxygenie, SLE 6000)

INTERVENTIONS:
Device: Closed-loop automated oxygen control (Oxygenie, SLE 6000) — The OxyGenie closed-loop oxygen saturation monitoring software (SLE) uses oxygen saturations from the SpO2 probe attached to the neonate, fed into an algorithm, to automatically adjust the percentage of inspired oxygen to maintain oxygen saturations within the target range. Manual adjustments including the percentage of FiO2 will be allowed at any point during the study if deemed appropriate by the clinical team.
  Arms: Closed-loop automated oxygen control

SUMMARY:
Many premature infants require respiratory support in the newborn period. Mechanical ventilation although life-saving is linked to complications for the lungs and other organs and its duration should be kept to a minimum. The use of supplemental oxygen may also increase the risk of comorbidities such as retinopathy of prematurity. Therefore, oxygen saturation levels and the amount of inspired oxygen concentration provided should be continuously monitored.

Oxygen control can be performed manually or with the use of a computer software incorporated into the ventilator that is called 'closed loop automated oxygen control'(CLAC). The software uses an algorithm that automatically adjusts the amount of inspired oxygen to maintain oxygen saturation levels in a target range. Evidence suggests that CLAC increases the time spent in the desired oxygen target range but there are no data to determine the effect on important clinical outcomes. A previous study has also demonstrated that CLAC reduces the inspired oxygen concentration more rapidly when compared to manual control. That could help infants come off the ventilator sooner.

With this study we want to compare the time preterm infants spend on the ventilator when we use the software to automatically monitor their oxygen levels with those infants whose oxygen is adjusted manually by the clinical team. That could help us understand if the use of automated oxygen control reduces the duration of mechanical ventilation and subsequently the complications related to it.

DETAILED DESCRIPTION:
This will be a randomised controlled trial. The investigators aim to recruit a minimum of seventy premature ventilated infants born at less than 31 weeks gestation. Participants will be randomised to either closed-loop automated oxygen control or manually controlled oxygen from recruitment to successful extubation. The investigators will also record basic epidemiologic parameters and associated comorbidities that may impact on the duration of mechanical ventilation. Infants with known congenital anomalies will be excluded from the study.

Informed written consent will be requested from the parents or legal guardians of the infants and the attending Neonatal Consultant will be requested to assent to the study.

Eligible infants whose parents consent to the study will be enrolled within 48 hours of initiation of mechanical ventilation.

Randomisation will be performed using an online randomisation generator. Patients will be ventilated using SLE6000 ventilators. Ventilation settings will be manually adjusted by the clinical team as per unit's protocol. The intervention group, in addition to standard care will be also connected to the OxyGenie closed-loop oxygen saturation monitoring software (SLE). This software uses oxygen saturations from the SpO2 probe attached to the neonate, fed into an algorithm, to automatically adjust the percentage of inspired oxygen to maintain oxygen saturations within the target range. Manual adjustments including the percentage of FiO2 will be allowed at any point during the study if deemed appropriate by the clinical team.

The nurse-to-patient ratio will be according to the unit's protocol that is determined on the patient's acuity.

Patients will be studied from enrolment until successful extubation. If an infant fails extubation and requires reintubation within 48 hours, he will be studied in his initial arm if less than 28 days old. Therefore, for those infants randomised at the intervention group CLAC will resume. Preterm infants that remain ventilated beyond day 28 of life will continue at their study arm (closed-loop automated oxygen control or manual oxygen control) till their first extubation attempt.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants less than 31 weeks completed gestation at birth requiring mechanical ventilation and admitted to King's NICU in the first 48 hours after birth

Exclusion Criteria:

* Preterm infants above 31 weeks completed gestation or term born infants
* Infants with major congenital abnormalities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-09-05 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
The duration of mechanical ventilation | Through study completion, an average of 2 years
  The duration of mechanical ventilation will be measured in median (interquartile range) number of days of ventilation for participants in each group.

SECONDARY OUTCOMES:
The percentage of time spent within target oxygen saturation range. | Through study completion, an average of 2 years
  Target oxygen saturation range for our preterm population is 90-95% as per local guideline. The time spent in target range will be calculated as a percentage of the total time of monitoring.
Number of manual adjustments to the inspired oxygen concentration required by clinical staff. | Through study completion, an average of 2 years
  The number of manual adjustment will be calculated by reviewing the infant's medical records.
Number of days on oxygen. | Through study completion, an average of 2 years
  The number of days each participant will require supplementary oxygen to maintain oxygen saturation levels within target range.
Length of Intensive Care stay | Through study completion, an average of 2 years
  The days each participant is admitted at the Neonatal Intensive Care
A diagnosis of bronchopulmonary dysplasia (BPD) at 36 weeks postmenstrual age | Through study completion, an average of 2 years
  The diagnosis of BPD will be calculated by reviewing the infant's medical records and respiratory status.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Greenough, Professor, Principal Investigator — King's College Hospital/ King's College London
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenough A. Long-term respiratory consequences of premature birth at less than 32 weeks of gestation. Early Hum Dev. 2013 Oct;89 Suppl 2:S25-7. doi: 10.1016/j.earlhumdev.2013.07.004. Epub 2013 Jul 30. PMID 23910576
- [Background] Di Fiore JM, Bloom JN, Orge F, Schutt A, Schluchter M, Cheruvu VK, Walsh M, Finer N, Martin RJ. A higher incidence of intermittent hypoxemic episodes is associated with severe retinopathy of prematurity. J Pediatr. 2010 Jul;157(1):69-73. doi: 10.1016/j.jpeds.2010.01.046. Epub 2010 Mar 20. PMID 20304417
- [Background] Hagadorn JI, Furey AM, Nghiem TH, Schmid CH, Phelps DL, Pillers DA, Cole CH; AVIOx Study Group. Achieved versus intended pulse oximeter saturation in infants born less than 28 weeks' gestation: the AVIOx study. Pediatrics. 2006 Oct;118(4):1574-82. doi: 10.1542/peds.2005-0413. PMID 17015549
- [Background] Ford SP, Leick-Rude MK, Meinert KA, Anderson B, Sheehan MB, Haney BM, Leeks SR, Simon SD, Jackson JK. Overcoming barriers to oxygen saturation targeting. Pediatrics. 2006 Nov;118 Suppl 2:S177-86. doi: 10.1542/peds.2006-0913P. PMID 17079621
- [Background] Sink DW, Hope SA, Hagadorn JI. Nurse:patient ratio and achievement of oxygen saturation goals in premature infants. Arch Dis Child Fetal Neonatal Ed. 2011 Mar;96(2):F93-8. doi: 10.1136/adc.2009.178616. Epub 2010 Oct 30. PMID 21037284
- [Background] Sturrock S, Ambulkar H, Williams EE, Sweeney S, Bednarczuk NF, Dassios T, Greenough A. A randomised crossover trial of closed loop automated oxygen control in preterm, ventilated infants. Acta Paediatr. 2021 Mar;110(3):833-837. doi: 10.1111/apa.15585. Epub 2020 Oct 6. PMID 32969040
- [Background] Sturrock S, Williams E, Dassios T, Greenough A. Closed loop automated oxygen control in neonates-A review. Acta Paediatr. 2020 May;109(5):914-922. doi: 10.1111/apa.15089. Epub 2019 Nov 27. PMID 31715041
- [Background] Dani C. Automated control of inspired oxygen (FiO2 ) in preterm infants: Literature review. Pediatr Pulmonol. 2019 Mar;54(3):358-363. doi: 10.1002/ppul.24238. Epub 2019 Jan 10. PMID 30632296
- [Background] Hunt KA, Dassios T, Ali K, Greenough A. Prediction of bronchopulmonary dysplasia development. Arch Dis Child Fetal Neonatal Ed. 2018 Nov;103(6):F598-F599. doi: 10.1136/archdischild-2018-315343. Epub 2018 Jun 12. No abstract available. PMID 29895571
- [Background] Dimitriou G, Greenough A, Endo A, Cherian S, Rafferty GF. Prediction of extubation failure in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2002 Jan;86(1):F32-5. doi: 10.1136/fn.86.1.f32. PMID 11815545
- [Background] Vliegenthart RJS, van Kaam AH, Aarnoudse-Moens CSH, van Wassenaer AG, Onland W. Duration of mechanical ventilation and neurodevelopment in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2019 Nov;104(6):F631-F635. doi: 10.1136/archdischild-2018-315993. Epub 2019 Mar 20. PMID 30894396
- [Derived] Kaltsogianni O, Dassios T, Jenkinson A, Jeffreys E, Ikeda K, Sugino M, Greenough A. Closed-loop automated oxygen control in preterm ventilated infants: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2025 Nov 10:fetalneonatal-2025-329022. doi: 10.1136/archdischild-2025-329022. Online ahead of print. PMID 41218846
- [Derived] Kaltsogianni O, Dassios T, Greenough A. Does closed-loop automated oxygen control reduce the duration of mechanical ventilation? A randomised controlled trial in ventilated preterm infants. Trials. 2022 Apr 8;23(1):276. doi: 10.1186/s13063-022-06222-y. PMID 35395952